CLINICAL TRIAL: NCT03803449
Title: Patient Satisfaction and Safety With Propofol Based Sedation With or Without Fentanyl for Gastrointestinal Endoscopy :a Prospective ,Randomized ,and Cohort Study
Brief Title: Patient Satisfaction and Safety With Propofol Based Sedation With or Without Fentanyl for Gastrointestinal Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Principal Investigator, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018SDU-QILU-069
Record Dates: First submitted 2018-04-22; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Patient Satisfaction
Keywords: propofol; fentanyl; gastrointestinal endoscopy
MeSH Terms: conditions — Patient Satisfaction | interventions — Propofol; Fentanyl; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to group A or B. Participants of group A are given propofol midazolam and fentanyl; while participants of group B are given propofol with midazolam without fentany
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Participants are given standard regimen: 50-200mg propofol and 1 mg midazolam
  Interventions: Drug: 50-200mg propofol; Drug: 1 mg midazolam
- Fentanyl group (Experimental): Participants are given intervention regimen: 50ug fentanyl, plus 50-200mg propofol and 1 mg midazolam.
  Interventions: Drug: 50-200mg propofol; Drug: 50ug fentanyl; Drug: 1 mg midazolam

INTERVENTIONS:
Drug: 50-200mg propofol — participants in both groups are given standard regimen including 50-200mg propofol.
  Other Names: Jingan, J20110055
Drug: 50ug fentanyl — participants in fentanyl group are given intervention regimen: 50ug fentanyl.
  Other Names: Yichang, H42022076
  Arms: Fentanyl group
Drug: 1 mg midazolam — participants in both groups are given standard regimen including 1 mg midazolam.
  Other Names: Liyuexi, H10980025

SUMMARY:
Patient satisfaction and safety with propofol based sedation with or without fentanyl for gastrointestinal endoscopy

DETAILED DESCRIPTION:
This study divide patients into two groups, one will be given propofol midazolam and fentanyl; another group was given propofol with midazolam without fentanyl; to observe two groups of patients blood pressure, body movement, and propofol dosage , and the difference in operator satisfaction, and how many people need to give fentanyl again; and two groups of patients after the operation of the reaction, if there are dizziness, nausea, and other adverse reactions; finally, the differences of these two schemes in different populations were analyzed, and the rationalization and individualized medication will be put forward.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patients scheduled for an outpatient gastrointestinal endoscopy by the principal investigator.

Exclusion Criteria:

* Patients with a history of colorectal surgery
* Patients with ASA class 4 or 5,
* Patients with pre-existing hypoxaemia (SpO2<90%),
* Patients with hypotension (SBP<90mmHg)
* Patients with bradycardia (HR<50 bpm)
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* patients with pregnancy or lactation
* Patients hemodynamically unstable
* Patients unable to give informed consent
* Patients with a history of drug allergies;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction assessed by the rate of vomit and diazzy after the procedure | half a year
  Rates of vomit and diazzy of patients after the procedure between the two groups

SECONDARY OUTCOMES:
Safety assessed by the rate of hypoxia during the procedure | half a year
  Hypoxia, defined as peripheral oxygen saturation <90% for >30 seconds
Safety assessed by the rate of hypotention during the procedure | half a year
  Hypotension, defined as systolic blood pressure <90 mmHg
Safety assessed by the rate of hyoxemia during the procedure | half a year
  Hypoxia, defined as peripheral oxygen saturation <90% for >30 seconds
Safety assessed by the rate of breadycardia during the procedure | half a year
  Bradycardia, defined as heart rate <50 beats/min
Safety assessed by the rate of required airway management during the procedure | half a year
  Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia
Safety assessed by the rate of involuntary movement during the procedure | half a year
  Involuntary movements, defined as unconscious movements requiring restraint or severe limb movement interrupting the endoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: yanqing li, Dr., Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Undecided